CLINICAL TRIAL: NCT07007078
Title: A Pilot Study to Evaluate the Therapeutic Effect of Dihydroartemisinin on Acne Vulgaris
Brief Title: Efficacy of Dihydroartemisinin for Treating Acne Vulgaris
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-113R
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; dihydroartemisinin
MeSH Terms: conditions — Acne Vulgaris | interventions — artenimol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DHA (dihydroartemisinin) Arm (Experimental)
  Interventions: Drug: dihydroartemisinin

INTERVENTIONS:
Drug: dihydroartemisinin — DHA 40mg tid for 90 days

SUMMARY:
The goal of this clinical trial is to learn if dihydroartemisinin (DHA) works to treat Acne Vulgaris in adults. The main question it aims to answer is:

• Does DHA improve the acne severity by at least one grade after treatment. Researchers will treat patients who are clinically diagnosed as Acne Vulgaris to see if DHA works to alleviate the symptoms of Acne Vulgaris.

Participants will:

* Take DHA every day for 3 months
* Visit the clinic once every month for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with acne vulgaris;
* For female patients, no pregnancy plans within the next 6 months.

Exclusion Criteria:

* Patients who have used sex hormones or other systemic medications for acne treatment within the past 3 months;
* Patients who have used topical medications for acne within the past 2 weeks;
* Pregnant or breastfeeding women;
* Patients with known severe diseases of vital organs (e.g., heart, liver, kidney) or malignancies.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of acne severity by Investigator's Global Assessment (IGA) | Before and immediately after 90-day treatment
  Improvement of acne severity is considered clinically significant if a subject's IGA improves by at least one grade

SECONDARY OUTCOMES:
Change of Global Acne Grading System (GAGS) score from baseline to the end of treatment | Before and immediately after 90-day treatment
  An improvement of ≥30% in the GAGS score will be considered significant
Change of inflammatory lesion count from baseline to the end of treatment | Before and immediately after 90-day treatment
Change of non-inflammatory lesion count from baseline to the end of treatment | Before and immediately after 90-day treatment
Number of participants who achieved an IGA score of 0 or 1 at the end of treatment | Before and immediately after 90-day treatment
Change of serum total testosterone from baseline to the end of treatment | Before and immediately after 90-day treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jingjing JIANG, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: After publication
Access Criteria: IPD and supporting information will be avaible to researchers upon reasonable request (e.g. with a practical and meaningful research proposal).